CLINICAL TRIAL: NCT04608695
Title: Ovarian Needle Puncture for Follicle Activation in IVF Patients With Diminished Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sezcan Mumusoglu, Associate Professor, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HU02
Record Dates: First submitted 2020-10-25; First posted 2020-10-29 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Activation of Primordial Follicles
Keywords: Follicle Activation; Premature Ovarian Insufficiency; Diminished Ovarian Reserve; Ovarian Puncture
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control ovary (No Intervention)
- Punctured ovary (Experimental)
  Interventions: Procedure: Ovarian puncture

INTERVENTIONS:
Procedure: Ovarian puncture — One side ovary of each patient included in the study, will be punctured 10 times under trans-vaginal ultrasound guidance with 17 gauge ovarian pick up needle, 1 month before the scheduled IVF cycle. Control group will be the other side ovary for each patient. Number of ≥ 14 mm follicle and collected oocytes will be compared.
  Arms: Punctured ovary

SUMMARY:
Premature ovarian insufficiency (POI), is cessation of ovarian function characterized by hypergonadotropic amenorrhea and hypoestrogenic syndrome before 40 years of age. About 1% of women younger than 40 years old and 0.1% before 30 are affected. POI imposes a great challenge on women's reproductive and long-term health, such as infertility, amenorrhea, osteoporosis, and cardiovascular disease. Most patients already had impaired or complete loss of fecundity when diagnosed. Currently, no optimal regimen exists to ameliorate ovarian function. Typically, they end up with egg donation or adoption as an alternative way. Less severe form of POI is diminished ovarian reserve (DOR). Although lack of consensus according to Bologna criteria cut off for DOR was defined as (antral follicle count (AFC) <5-7 follicles or anti-Mullerian hormone (AMH) <0.5-1.1 ng/ml).

Previously it has been showed that 24% of women with POI had resumption of ovarian function and 4% resulted in baby births. These data indicates residual follicles are available in atrophic ovaries and have potential for development and even fertilization. In routine IVF practice 15% percent of patients have poor ovarian response to ovarian stimulation. Patients with DOR with a previous poor ovarian response (cycles cancelled or yielding ≤3 oocytes with a conventional protocol) might have benefit from the strategies increasing follicle activation and number of growing follicles and oocyte retrieved. Therefore, strategies enabling ovarian resumption predictable and follicle activation feasible are promising for POI/DOR treatment. Recently, In vitro Activation (IVA) approach has been proposed and live births have been achieved in patients with POI. Phosphatase and tensin homolog (PTEN) enzyme inhibitors and phosphatidylinositol-3 kinase activators could activate AKT pathway and activate the dormant follicles. Ovarian fragmentation could lead to ovarian primary follicle growth by interfering with Hippo signaling pathway. Residual follicles in patients with POI could be activated to develop for egg retrieval by combination of mechanical and chemical stimulation.

In 2019, Zhang et al retrospectively analyzed the follicle development and pregnancy outcome in 80 POI patients after laparoscopic ovarian biopsy/scratch without using chemical agents as was the case in IVA. 11 (13.75%) patients presented with ovarian function resumption, three metaphases II oocytes were retrieved in 10 patients and two embryos were formed and freshly transferred followed by a healthy singleton delivery in 1 (1.25%) patient. They concluded that the technique of ovarian biopsy/scratch without chemical activation could promote follicle development in vivo, suggesting it could bring promising benefits for some women with POI.

In patient with POI/DOR, activation of residual follicles is a promising option and further studies are warranted. Previous studies included laparoscopic surgery which may lead to possible surgical complications. Without using chemical agents and laparoscopic surgery, main object of this study is mechanical follicle activation with trans-vaginal ovarian needle puncture with 17 gauge oocyte pickup needle in IVF patients with DOR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diminished ovarian reserve
* <3 oocytes collected in previous cycle (with anti-mullerian hormone <0.5 ng/mL and/or antral follicle count <5)
* Cycles stimulated with flexible antagonist protocol
* Cycles triggered with recombinant hCG
* Fresh transfer cycles
* Patients with <40 years of age
* BMI <30 kg/m2

Exclusion Criteria:

* Preimplantation genetic testing
* Azospermia

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of ≥14 mm follicle | 4 month after intervention as a response to ovarian stimulation
  Number of ≥14 mm follicle on the trigger day
Antral follicle count | 4 month after intervention on the second/third day of menstrual cycle
  Antral follicle count

SECONDARY OUTCOMES:
Number of collected oocytes | 4 month after intervention as a response to ovarian stimulation
  Number of collected oocytes on the oocyte pick-up day

CONTACTS AND LOCATIONS:
Overall Officials: Sezcan Mumusoğlu, Assoc. Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe UniversityHacettepe University School of Medicine, Department of Ob/Gyn, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] De Vos M, Devroey P, Fauser BC. Primary ovarian insufficiency. Lancet. 2010 Sep 11;376(9744):911-21. doi: 10.1016/S0140-6736(10)60355-8. Epub 2010 Aug 11. PMID 20708256
- [Background] Torrealday S, Kodaman P, Pal L. Premature Ovarian Insufficiency - an update on recent advances in understanding and management. F1000Res. 2017 Nov 29;6:2069. doi: 10.12688/f1000research.11948.1. eCollection 2017. PMID 29225794
- [Background] Ferraretti AP, Gianaroli L. The Bologna criteria for the definition of poor ovarian responders: is there a need for revision? Hum Reprod. 2014 Sep;29(9):1842-5. doi: 10.1093/humrep/deu139. Epub 2014 Jul 9. PMID 25008235
- [Background] Bachelot A, Nicolas C, Bidet M, Dulon J, Leban M, Golmard JL, Polak M, Touraine P. Long-term outcome of ovarian function in women with intermittent premature ovarian insufficiency. Clin Endocrinol (Oxf). 2017 Feb;86(2):223-228. doi: 10.1111/cen.13105. Epub 2016 Jun 14. PMID 27177971
- [Background] Chen X, Chen SL, Ye DS, Liu YD, He YX, Tian XL, Xu LJ, Tao T. Retrospective analysis of reproductive outcomes in women with primary ovarian insufficiency showing intermittent follicular development. Reprod Biomed Online. 2016 Apr;32(4):427-33. doi: 10.1016/j.rbmo.2015.12.011. Epub 2016 Jan 14. PMID 26825246
- [Background] Kawamura K, Kawamura N, Hsueh AJ. Activation of dormant follicles: a new treatment for premature ovarian failure? Curr Opin Obstet Gynecol. 2016 Jun;28(3):217-22. doi: 10.1097/GCO.0000000000000268. PMID 27022685
- [Background] Zhang X, Han T, Yan L, Jiao X, Qin Y, Chen ZJ. Resumption of Ovarian Function After Ovarian Biopsy/Scratch in Patients With Premature Ovarian Insufficiency. Reprod Sci. 2019 Feb;26(2):207-213. doi: 10.1177/1933719118818906. Epub 2018 Dec 12. PMID 30541396